CLINICAL TRIAL: NCT01129622
Title: Phase II Study of the Effect of Acute Aromatase Inhibition on Breast MRI Postmenopausal Women
Brief Title: Effect of Aromatase Inhibitors on Breast Magnetic Resonance Imaging (MRI)
Acronym: RFCLET2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Robert Casper, Professor, Obstetrics and Gynecology, Mount Sinai Hospital, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CFWH-AI1
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer
Keywords: Letrozole; Breast MRI; Postmenopausal women
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Letrozole, Breast enhancement, Safety (Experimental): Single arm of healthy postmenopausal women who received baseline diagnostic MRI will receive letrozole of 12.5 mg/day orally for three successive days. A second post treatment breast MRI is done right after receiving the three days of letrozole treatment and within one month after the first MRI .
  Interventions: Drug: letrozole

INTERVENTIONS:
Drug: letrozole — Letrozole (12.5 mg/day ) which is higher than the dose routinely used for therapeutic indications is given for a brief duration (3 successive days) aiming to promote acute aromatase inhibition suitable for pre-diagnostic regimens.
  Other Names: Femara TM Novartis Pharmaceuticals Canada Inc., Dorval, QC

SUMMARY:
This study is a primary investigation to determine the usefulness and safety of a short course of a relatively high dose of letrozole (a medication used to decrease the female hormone estrogen which is produced locally inside the breast after menopause) in improving the performance of of breast MRI (Magnetic Resonance Imaging). The inhibition of estrogen in the breast by letrozole might help better identifying of suspicious areas in the breast and could assist radiologists in distinguishing between benign breast areas and cancer tissue. This might help reducing the rate of call backs and unnecessary biopsies for patients. We expect to enroll 20 healthy postmenopausal women in this study.

DETAILED DESCRIPTION:
A breast MRI will be performed in the standard way for diagnosis and to serve as a baseline. A second MRI will be performed within a month and following administration of letrozole 12.5 mg daily for three days to reduce breast estrogen levels and in anticipation of lowering breast gadolinium dye uptake.

ELIGIBILITY:
Inclusion Criteria:

* Women are eligible to participate if they are 40 years or older and have been menopausal (had no menstrual bleeding during the past 12 months)

Exclusion Criteria:

* History of bilateral mastectomy, osteoporosis or renal impairment.

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Casper, MD, Principal Investigator — Mount Sinai Hopsital
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Result] Mousa NA, Eiada R, Crystal P, Nayot D, Casper RF. The effect of acute aromatase inhibition on breast parenchymal enhancement in magnetic resonance imaging: a prospective pilot clinical trial. Menopause. 2012 Apr;19(4):420-5. doi: 10.1097/gme.0b013e31823772a8. PMID 22258545

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 women over age 40 on hormone therapy were recruited. No previous abnormal breast imaging.
Groups:
- Letrozole, Breast Enhancement, Safety: Single arm of healthy postmenopausal women to have two breast MRI (baseline and post-treatment). Letrozole of 12.5 mg/day is given for three successive days just prior to the second MRI.
Period: Overall Study
Arm/Group | Letrozole, Breast Enhancement, Safety
Started | 16
Completed | 14
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Letrozole, Breast Enhancement, Safety
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Region of Enrollment [Number; unit: participants]
  Canada | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Women With Reduced Breast Parenchymal Enhancement
Description: Image analysis was done using the e-film workstation. A region of interest was selected in all images. The signal intensity of enhancement was recorded and the relative enhancement (percentage of increase in signal intensity) was calculated as (SIc - SI)/SI × 100, where SI and SIc are the precontrast and the postcontrast signal intensities, respectively. Relative enhancement was compared at the baseline MRI study and the after one month MRI study for all participants.
Time Frame: One month MRI study after letrozole compared to baseline MRI study, both with gadolinium enhancement
Population: All participants who completed two MRIs were analysed. Percentage reduction in breast enhancement compared to baseline was determined.
Measure: Number; unit: Number of participants
Arm/Group | Letrozole, Breast Enhancement, Safety
Number analyzed (Participants) | 14
Number of participants | 7

2. Secondary Outcome: Number of Participants Developed Adverse Effects of 12.5 mg of Letrozole
Description: The number of participants who developed short term hypoestrogenic side effects or other adverse effects of letrozole during the intake of the medication or in the following week.
Time Frame: Three days plus One Week following medication
Population: All entered subjects
Measure: Number; unit: Number of participants
Groups:
- Adverse Events: Hypo-estrogenic side effects
Arm/Group | Adverse Events
Number analyzed (Participants) | 14
Number of participants | 3

ADVERSE EVENTS:
Time Frame: 10 months
Description: Subject report of adverse events prior to second MRI.
Arm/Group | Letrozole, Breast Enhancement, Safety
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole, Breast Enhancement, Safety (N=14)
Headache (Nervous system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 — Mild arthralgia

LIMITATIONS AND CAVEATS:
The small sample size is a limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No